CLINICAL TRIAL: NCT06353919
Title: Remotely-delivered Yoga Nidra for Decreasing Use of BZRAs for Insomnia and Anxiety in Older Adults
Brief Title: Remote Yoga Nidra for Deprescribing BZRAs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ryan Bradley, Director, Helfgott Research Institute, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NUNM
Record Dates: First submitted 2023-11-14; First posted 2024-04-09 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Anxiety; Insomnia
Keywords: Yoga; Anxiety; Insomnia; Benzodiazepine
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Nidra (Experimental): Participants will practice 30 minutes of yoga nidra 3-5x's/week for 6 weeks
  Interventions: Other: Yoga Nidra
- Sleep Hygiene, Anxiety, and Benzodiazepine Receptor Agonist Education (Active Comparator): Participants will review education material for 30 minutes at a time, 3-5x's/week for 6 weeks
  Interventions: Other: Sleep Hygiene, Anxiety, and Benzodiazepine Receptor Agonist Education

INTERVENTIONS:
Other: Yoga Nidra — Recordings were created to allow participants access to a variety of Yoga Nidra practices. Participants will be instructed to complete a 30-minute Yoga Nidra 3-5 times per week, at any time of day or night (including before bed and/or during bouts of sleeplessness). This duration and frequency is informed by previous studies.
  Related to intentionally decreasing BZRA use, the recording requests each practitioner to set a resolve/personal goal at the start of each practice, and they are asked to repeat it again at the end. In our study, participants will be asked to develop a short and simple resolve in their own words, related to reducing BZRA use, improving sleep and decreasing anxiety, and they will be asked to recite it at each practice.
  Arms: Yoga Nidra
Other: Sleep Hygiene, Anxiety, and Benzodiazepine Receptor Agonist Education — Participants will be instructed to access excerpts from standardized and trusted materials through our online platform for 30 minutes, 3-5 times per week.
  Arms: Sleep Hygiene, Anxiety, and Benzodiazepine Receptor Agonist Education

SUMMARY:
The overall goal of this application is to assess feasibility and impact of a remotely delivered guided meditation practice called Yoga Nidra, for reducing or stopping use of Benzodiazepine Receptor Agonists (BZRAs) for insomnia and anxiety in a population of older adults recruited from within the Birmingham VA medical system.

DETAILED DESCRIPTION:
Before 2020, insomnia and anxiety were estimated to affect much of the US adult population at some point in their life (50% and 30% respectively). By summer of 2022, however, daily negative impacts of insomnia and anxiety were reported by 28% and 52% of US adults, respectively. In the absence of intervention, the COVID-19 pandemic will have lasting negative impacts on our society's sleep and mental health, plus contribute to increased mortality due to depression, heart disease and stroke resulting from insomnia and anxiety. Insomnia and anxiety often co-exist and generalized anxiety disorder is the most common co-morbid psychiatric condition diagnosed with insomnia, with 73% of individuals suffering from anxiety later developing insomnia. Although Benzodiazepine Receptor Agonists (BZRAs) provide rapid symptom relief, they carry risks of side effects including addictive potential, greater risk for falls and motor vehicle accidents, and potential respiratory failure resulting in death, especially when combined with other CNS suppressants such as opiates. Furthermore, many medications may require life-long use, and long-term safety and efficacy have not been established, plus cost remains a barrier to access and adherence. As a result, the first-line treatment for insomnia and anxiety is often Cognitive Behavioral Therapy (CBT). However, CBT is difficult to access, expensive, and takes 4-6 weeks before clinical benefit becomes evident. And it is not very effective in eliminating long-term BZRA use [18] or insomnia/anxiety (34% remission rate for individuals with insomnia and comorbid anxiety). Thus, there is need to test accessible, fast-acting therapies, as stand-alone treatments, or precursor therapies in a stepped care model with CBT-I, to decrease BZRAs used for insomnia and anxiety.

Mind-body therapies offer one solution as they are purported to increase self-efficacy and self-regulation, potentially helping to facilitate cognitive and behavioral change needed to decrease BZRA use, and to modify sleep and anxious thought patterns. Importantly, for individuals who struggle to fall asleep or stay asleep (often resulting when anxiety exists alongside insomnia) a fast-acting therapy needs to be accessible in the middle of the night. An effective mind-body therapy for comorbid insomnia and anxiety requires specific qualities such as ease of access, ease of adoption, and mechanisms that support sleep such as inducing relaxation.

Remotely-delivered interventions for insomnia and anxiety have been in greater demand since healthcare systems became strained by the pandemic. They offer a valuable opportunity for easy access, and there is evidence of effectiveness. Yet there remains room for improvement, and there has been limited research on remotely-delivered mind-body interventions. Yoga Nidra, a remotely-delivered 30-minute guided meditation (practiced by listening to a voice, while lying down with eyes closed) could be an excellent practice to address insomnia as it is relaxing, free, easily accessible, and only requires passive involvement. It naturally produces a hypnogogic state, which occurs during a normal transition to sleep and promotes a state of deep rest (with simultaneous release of physical, mental, and emotional tensions), accompanied by a unique change in awareness, allowing passive self-exploration, resolution, and growth. The practice is described in detail elsewhere, and is scripted, making it easily reproducible for research, clinical, and personal use. Importantly, this practice can be used at any time of day or night (including to help fall asleep) and requires no special physical capabilities or movements. Setting it apart from BZRAs or CBT-I, Yoga Nidra has no limitations for long-term use (such as side effects or cost) and in fact, ongoing practice provides regular opportunities for self-exploration and biopsychosocial benefit.

Relevance to Deprescribing in Older Adults: In spring of 2021, 32% of older adults had reported increased sleep disturbances since the start of the pandemic, and amongst those individuals 78% reported "trouble falling or staying asleep". Additionally, with 44% of older adults reporting self-medicating when they could not sleep, especially since COVID-19 began, risks must be considered. Further complicating matters, issues of polypharmacy and cognitive decline, make safe BZRA use more difficult to ensure in older adults. With 20-30% of older adults suffering daily from anxiety and insomnia, Yoga Nidra is a very promising, accessible, passive, low-cost, and rapid-acting intervention to turn to, instead of BZRAs, for help falling asleep, improving sleep quality, and decreasing anxiety. Yoga Nidra could be especially helpful to those with hypnotic-dependent insomnia, as it is traditionally used to break habits and addictions, with reports of practitioners spontaneously quitting smoking or drinking. This phenomenon was also observed in our work and is attributed to deeply tuning in to what is best for oneself. Description of the Population to be Served: This study will focus on adults in the US over age 65, who are using BZRAs for insomnia comorbid with anxiety, have been using them regularly for at least 3 months, and who are interested in decreasing or discontinuing usage.

ELIGIBILITY:
Inclusion Criteria:

* over 65 years of age
* Use of benzodiazepine receptor agonist medication at least 3 nights per week for a minimum of three months and wish to decrease their use
* Ability to speak, read, and understand English
* Ability to sit or lie comfortably for 30 minutes at a time
* Must be under the care of a primary care provider

Exclusion Criteria:

* current use of sleep or anxiety medication other than benzodiazepine receptor agonists
* severe depression as indicated by a score above 20 on the patient health questionnaire
* presence of other comorbidities that may impact sleep i.e. restless leg syndrome, narcolepsy, or others)
* regular mind/body practice within 6 months
* unavoidable lifestyle disruptions to sleep

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Demand | Up to one year
  Number of inquiries
Recruitment Success | Up to one year
  Whether 30 participants will enroll and complete the 6-week study
Implementation practicality | Up to one year
  Whether the interventions can be successfully administered remotely in this population
Acceptability | 6 weeks
  Comfort and tolerability ratings on a 0-100 scale
Retention | 6 weeks
  Attrition Rate
Adherence to Protocol | 6 weeks
  Percentage of participants who adhered to each intervention

SECONDARY OUTCOMES:
Use of Benzodiazepine Receptor Agonist medications | 6 weeks
  Frequency and amount used during the study
Cessation of Benzodiazepine Receptor Agonist medication | 6 weeks
  Number of participants not taking Benzodiazepine medication by the end of the trial
Baseline Urine Benzodiazepine Receptor Agonist Concentration | Baseline
  Concentration of Benzodiazepine metabolites in urine
Close-out Urine Benzodiazepine Receptor Agonist Concentration | Week 6
  Concentration of Benzodiazepine metabolites in urine

OTHER OUTCOMES:
Insomnia Severity Index | Baseline
  Validated measure of insomnia severity
Insomnia Severity Index | Week 6
  Validated measure of insomnia severity
Insomnia Severity Index | Month 1
  Validated measure of insomnia severity
Insomnia Severity Index | Month 3
  Validated measure of insomnia severity
Patient reported outcomes measurement information system 29 | Baseline
  Self reported assessment of sleep quality, pain, and anxiety
Patient reported outcomes measurement information system 29 | Week 6
  Self reported assessment of sleep quality, pain, and anxiety
Generalized Anxiety Disorder 7 Questionnaire | Baseline
  Average GAD7 score
Generalized Anxiety Disorder 7 Questionnaire | Week 6
  Average GAD7 score

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, ND,MPH, Principal Investigator — National University of Natural Medicine